CLINICAL TRIAL: NCT04720378
Title: A Phase 1, Multi-Center, Open-Label, Safety and Tolerability Study of Intravenous Administration of ST266 in Subjects With Confirmed COVID-19 Infection
Brief Title: Safety and Tolerability Study of IV ST266 in COVID-19 Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Noveome Biotherapeutics, formerly Stemnion (Industry)
Collaborators: IQVIA Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ST266-CRS-101
Record Dates: First submitted 2021-01-21; First posted 2021-01-22 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Cytokine Release Syndrome
Keywords: COVID-19
MeSH Terms: conditions — Cytokine Release Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): 0.1 ml/kg IV ST266 once a day for 5 days
  Interventions: Biological: ST266
- Cohort 2 (Experimental): 0.25 ml/kg IV ST266 once a day for 5 days
  Interventions: Biological: ST266
- Cohort 3 (Experimental): 0.5 ml/kg IV ST266 once a day for 5 days
  Interventions: Biological: ST266
- Cohort 4 (Experimental): 1.0 ml/kg IV ST266 once a day for 5 days
  Interventions: Biological: ST266

INTERVENTIONS:
Biological: ST266 — 1X ST266

SUMMARY:
The primary aim of the study is to evaluate the safety and tolerability of open-label ST266 given to subjects with confirmed COVID-19 infection through IV administration once a day of 5 consecutive days.

DETAILED DESCRIPTION:
This clinical trial will utilize a 3+3 enrollment design with sentinel approach.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant/non-breastfeeding females age 18-70 years of age.
2. Laboratory confirmed SARS-CoV-2 infection determined by PCR or other commercial/public health assay (test results must be obtained within 7-days of the Screening Visit).
3. BMI between 18 and 39 inclusive, with a maximum weight of 150 kg (330lbs).
4. Asymptomatic or mildly symptomatic COVID-19 positive subject with a score of 1 or 2 on the WHO 7-point ordinal scale.
5. Subjects with pulse oximetry of > 94% on room air
6. Subjects have controlled blood pressure of < 160/100 mmHg or systolic BP > 90 mmHg (or 20 mmHg less than usual range, whichever is higher)
7. Subjects with pulse < 120 bpm
8. Willingness and ability to comply with study-related procedures and assessments.
9. If female, subjects must use an effective method of birth control or abstain from sexual relations with a male partner (unless has undergone tubal ligation or is 1 year postmenopausal) for their duration of study participation.
10. If male, subjects must use an effective method of birth control or abstain from sexual relations with a female partner (unless has undergone a vasectomy and it has been more than 6 months) for their duration of study participation.
11. Subject or subject's legal representative provides written consent prior to the initiation of any Screening or study specific procedures.

Exclusion Criteria:

1. Subjects requiring immediate admission to the hospital due to complications of COVID-19 infection.
2. Subject has an untreated active bacterial, fungal, viral or other infection not related to COVID-19 infection.
3. Subjects with chronic lung diseases of any etiology including idiopathic pulmonary fibrosis, Tuberculosis, COPD, persistent asthma, and pulmonary hypertension.
4. Subjects with a severe history of cardiac disease (such as congestive heart failure, coronary artery disease, cardiac arrhythmia)
5. Subjects with a history of neurological disorders (such as epilepsy, stroke, encephalopathy, Guillain-Barré syndrome)
6. Subjects with D-dimer > 2 ug/mL
7. Subjects with a history of coagulopathy or currently taking anti-coagulation medication
8. Subjects with PTT ≥ 100s or INR ≥ 2.75
9. Malignancy in the last 5 years (except successfully treated basal cell carcinoma).
10. Stage 4 severe chronic kidney disease or requiring dialysis (i.e., eGFR < 30).
11. Subjects with a reactive or positive screening test result For Hepatitis A virus immunoglobulin M (HAV IgM), Hepatitis B Surface Antigen (HBsAg), Hepatitis C Virus Antibody (HCVAb) or Human Immunodeficiency Virus Antibody (HIVAb).
12. TBIL> 2×ULN, ALT > 3×ULN, AST> 3×ULN, or ALP> 3×ULN.
13. Neutrophils <1000/mm3, PLT<50×10^9/L, or HGB<8g/dL
14. Previous participation in any other interventional clinical trial for the treatment for COVID-19.
15. Subject actively participating in any other clinical study (with the exception of observational studies where there is no intervention with an investigational product or device)
16. Use of anti-cancer or immunomodulatory biological drug or kinase inhibitor (e.g., tocilizumab, sarilumab) or, JAK inhibitors (within 30 days of enrollment or five times the half-life [whichever is longer]).
17. Chronic glucocorticosteroid use equivalent to daily oral prednisone > 10 mg per day (10 mg oral prednisone every other day is allowed).
18. Live (live-attenuated) vaccines are not permitted within 2 weeks prior to enrollment or during the study treatment and safety follow-up periods, including the SARS-CoV-2 vaccine (with the exception of the Flu vaccine which is allowed at any time)
19. Subject is pregnant or breastfeeding or plans to become pregnant within 12 months.
20. Subjects with a history of alcohol or drug abuse, or the use of illicit drugs within the 12 months prior to Screening or use of medical marijuana within 1 month prior to Screening.
21. Subject is considered by the Investigator, for any reason, to be an unsuitable candidate for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Treatment-Emergent Adverse Events | 3 months
  Determine the incidence and severity of treatment-emergent adverse events related to the IV administration of ST266 based on findings from physical examinations, laboratory evaluations, vital signs, and ECG measurements.

SECONDARY OUTCOMES:
Pulse Oximetry | 14 days
  Percent improvement in pulse oximetry from Baseline to Day 14
Fever | 14 days
  Time to resolution of fever
Clinical Status on Ordinal Scale | 14 days
  Improvement or absence of worsening in clinical status on WHO 7-point ordinal scale from baseline to Day 14

OTHER OUTCOMES:
TNFα at Day 6 | 6 days
  Change in TNFα from Baseline through Day 6
IL- 1β at Day 6 | 6 days
  Change in IL- 1β from Baseline through Day 6
IL-6 at Day 6 | 6 days
  Change in IL-6 from Baseline through Day 6
TNFα at Day 14 | 14 days
  Change in TNFα from Baseline through Day 14
IL- 1β at Day 14 | 14 days
  Change in IL- 1β from Baseline through Day 14
IL-6 at Day 14 | 14 days
  Change in IL-6 from Baseline through Day 14

CONTACTS AND LOCATIONS:
Overall Officials: David L Steed, MD, Study Director — Noveome Biotherapeutics, Inc
Locations (3):
- United States (3):
  - Innovative Research of West Florida, Clearwater, Florida
  - Great Lakes Clinical Trials, Chicago, Illinois
  - WR-ClinSearch, LLC, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No